CLINICAL TRIAL: NCT01899183
Title: Effectiveness of Anti-reflux Surgery for the Cure of Chronic Cough Associated With Gastro-oesophageal Reflux Disease
Brief Title: Surgery in Chronic Cough GERD Related
Acronym: CCGERD
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: Chronic Cough and GERD
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: GERD
Keywords: Chronic cough; Esophagus; Gastro-esophageal reflux disease; Esophageal surgery; Minimally invasive surgery; Extra-esophageal reflux symptoms.
MeSH Terms: conditions — Gastroesophageal Reflux; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Anti-reflux Surgery — Nissen Fundoplication; Collis Gastroplasty

SUMMARY:
The effectiveness of surgical fundoplication in treating classical reflux symptoms is well documented, but the role of surgery in alleviating extra-esophageal symptoms allegedly secondary to gastro-esophageal reflux disease (GORD) is far to be assessed.

The effectiveness of anti-reflux surgery on extra-esophageal reflux symptoms varies from 15% to 95%; the spread of these data is largely attributable to disparate study design and methodology, patient selection, and outcome metrics.

In order to assess whether anti-reflux surgery may have beneficial effects on chronic cough allegedly secondary to GERD and to eventually identify the preoperative clinical profile which could predict those positive effects, we considered two groups of patients presenting with 1) GERD associated to chronic cough, 2), typical GERD who underwent anti-reflux surgery.

DETAILED DESCRIPTION:
Pre-operatively, patients routinely underwent the symptoms assessment, barium swallow, upper gastro-intestinal endoscopy and esophageal manometry.

The type and severity of symptoms and the grade of reflux oesophagitis were scored using a questionnaire with semi-quantitative scales.

The upper gastro-intestinal (GI) endoscopy, barium swallow and esophageal manometry were performed according to standard techniques; reflux esophagitis was reported according to the Los Angeles classification. In the absence of Los Angeles grade A or higher esophagitis, patient underwent a 24h pH-recording or intraluminal impedance/pH monitoring. Patients complaining of chronic cough were submitted to a specific work-up consisting of a chest High Resolution Computed Tomography (HRCT) scan, methacholine challenge test and spirometry in order to exclude pulmonary diseases.

Surgery was performed in patients negative for pulmonary diseases on chest HRCT scan, on methacholine challenge test and spirometry, in consideration of the fact that patients had been referred mainly for the therapy of chronic cough.

The study was started in 1995 and it was closed in 2010.

ELIGIBILITY:
Inclusion Criteria:

patients aged > 18 years, affected by chronic cough (> 8 weeks)associated with GERD typical symptoms, negative for pulmonary diseases on chest HRCT scan, on methacholine challenge test and spirometry, undergoing anti-reflux surgery

Exclusion Criteria:

patients with chronic cough (> 8 weeks) positive for pulmonary diseases on chest High Resolution Computed Tomography (HRCT) scan, methacholine challenge test and spirometry; association of GERD with epiphrenic esophageal diverticulum, collagen diseases, undetermined esophageal motility disorders, redo antireflux surgery, previous surgery on the thoracic and abdominal esophagus and stomach,on the diaphragm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GERD and Chronic Cough (< 8 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 1995-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Global Results and Resolution of chronic cough | minimum 12 months
  Pre-operatively, patients routinely underwent the symptoms assessment, barium swallow, upper gastro-intestinal endoscopy, esophageal manometry, chest High Resolution Computed Tomography scan, methacholine challenge test and spirometry. Surgery was performed on patients positive for gastro-esophageal reflux disease and negative for pulmonary diseases.
  The type and severity of symptoms and the grade of reflux esophagitis were scored using a questionnaire with semi-quantitative scales (form 0 = absence of symptoms or esophagitis, to 3 = severe symptoms and esophagitis.For the surgical results an evaluation scale , from "excellent" to "poor", was used.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, MD, Principal Investigator — Departement of Medical and Surgical Sciences University of Bologna
Locations (1):
- Department of Medical And Surgical Sciences University of Bologna, Bologna, BO, Italy

REFERENCES:
- See also: Department of Medical and Surgical Sciences University of Bologna — http://www.dimec.unibo.it/it